CLINICAL TRIAL: NCT01064089
Title: A Phase I Dose Escalation, Multi-center, Open-label Study of HSP990 Administered Orally Once Weekly in Adult Japanese and Korea Patients With Advanced Solid Malignancies
Brief Title: Dose Escalation of HSP990 in Japan/Korea
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHSP990A1101
Record Dates: First submitted 2010-02-01; First posted 2010-02-08 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2012-12

CONDITIONS: Advanced Solid Tumors
Keywords: HSP990; HSP90; Japan/Korea; Phase I; advanced solid tumors; dose escalation; maximum tolerated dose; MTD; Japanese paatients; Korean patients
MeSH Terms: interventions — 2-amino-7-(4-fluoro-2-(6-methoxypyridin-2-yl)phenyl)-4-methyl-7,8-dihydropyrido(4,3-d)pyrimidin-5(6H)-one

ARMS (1):
- HSP990 (Experimental): dose escalation
  Interventions: Drug: HSP990

INTERVENTIONS:
Drug: HSP990

SUMMARY:
This study is a phase I dose escalation, multi-center, open-label study of HSP990 administered orally once weekly in adult Japanese and Korea patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced solid tumors (advanced cancer)
2. Patient's disease must be evaluable using the RECIST criteria
3. Patients must be 18 or older in Korea or 20 or older in Japan
4. Patients must be relatively healthy as measured by their performance status
5. Patients must have acceptable laboratory values as measured by blood tests
6. Patients must be able to swallow capsules
7. Patients must understand the study and give written permission to enter study

Exclusion Criteria:

1. Patients cannot have brain tumors
2. Patients cannot have had prior medicines that are similar to the study drug or an HDAC inhibitor medicine
3. Patients must not be classified as a "poor or intermediate CYP2C9 metabolizer" as measured using a sample of their blood
4. Patients must have recovered from all previous anti-cancer therapy
5. Patients must have finished taking their previous anti-cancer therapy before entering study
6. Patients must not have a severe disease at the time of study entry (for example: severe diarrhea, disease of the liver or kidney, other cancers, etc.)
7. Patients must have relatively good heart function

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
establish maximum tolerated dose (MTD) | 2.5 years

SECONDARY OUTCOMES:
Safety by measuring occurrence of dose limiting toxicity (DLT) and other adverse events | 2.5 years
Efficacy by collecting data on response (complete response [CR], partial response [PR]) and stable disease (SD) | 2.5 years
Establishment of a pharmacokinetic profile by collecting information on parameters including but not limited to Cmax, Tmax, T1/2 and AUC in plasma samples | 2.5 years
Measurement of biomarkers for HSP90 pathway in blood and tissue | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba

REFERENCES:
- See also: Results for CHSP990A1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7623